CLINICAL TRIAL: NCT02492893
Title: Yoga Intervention for Substance Use and Antiretroviral Therapy Adherence in Community
Brief Title: Yoga Intervention for Substance Use and ART Adherence in Community Reentry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Peter McManus Charitable Trust (Other); National Coalition of Independent Scholars (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 820294; 1F31DA038429-01 (NIH)
Record Dates: First submitted 2015-06-19; First posted 2015-07-09 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Substance Related Disorders; HIV
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hatha Yoga (Experimental): A 12-session 90-minute weekly hatha yoga intervention, that includes asanas (physical postures), pranayama (breathing exercises) and dhyana (meditation.
  Interventions: Other: Hatha yoga
- Treatment as Usual (No Intervention)

INTERVENTIONS:
Other: Hatha yoga
  Arms: Hatha Yoga

SUMMARY:
People with HIV and a substance use disorder who are reentering the community from prison or jail face the dual risks of relapse and interruptions in adherence to antiretroviral therapy (ART) medication. This mixed-methods randomized controlled trial will compare the stress, substance use and ART adherence outcomes of participants in a 12-session, 90-minute weekly yoga group intervention with participants in a treatment as usual control group. All participants are re-entering the community, have HIV and experience substance use challenges.

ELIGIBILITY:
Inclusion Criteria:

* have HIV
* experience substance use challenges, within one year of reentry from prison or jail

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2014-12; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Stress: Perceived Stress Scale (self-report) | 3 months
Substance use: Time Line Follow Back (self-report) | 3 months

SECONDARY OUTCOMES:
Antiretroviral therapy adherence: prescription refill (pharmacy data) | 3 months
Heart rate: sphygmomanometer | 3 months
Blood pressure: sphygmomanometer | 3 months
Viral load: blood test | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States